CLINICAL TRIAL: NCT04115878
Title: Evaluation of Atomoxetine and Oxybutynin for Obstructive Sleep Apnea in Children With Down Syndrome
Brief Title: Medications for Obstructive Sleep Apnea In Children With Down Syndrome
Acronym: MOSAIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Daniel A. Combs, Assistant Professor of Pediatrics, University of Arizona
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1908864846; R61HL151254 (NIH)
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Obstructive Sleep Apnea; Down Syndrome
Keywords: atomoxetine; oxybutynin
MeSH Terms: conditions — Sleep Apnea, Obstructive; Down Syndrome | interventions — Atomoxetine Hydrochloride; oxybutynin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- High dose ato-oxy (Active Comparator)
  Interventions: Drug: Atomoxetine and oxybutynin (ato-oxy)
- Low dose ato-oxy (Active Comparator)
  Interventions: Drug: Atomoxetine and oxybutynin (ato-oxy)

INTERVENTIONS:
Drug: Atomoxetine and oxybutynin (ato-oxy) — Low dose ato-oxy will include 0.5 mg/kg/day of atomoxetine (max 40 mg) in combination with 5 mg oxybutynin High dose ato-oxy will include 1.2 mg/kg/day atomoxetine (max 80 mg) and 5 mg oxybutynin

SUMMARY:
This is a randomized, double blind, cross-over study of the combination of atomoxetine and oxybutynin (ato-oxy) in children with DS and OSA documented by polysomnography (PSG). Participants will receive high dose ato-oxy for four weeks as well as low dose ato-oxy for four weeks in random order. During the high dose ato-oxy period, participants will take 5 mg oxybutynin and 0.5mg/kg/day (max 40 mg) atomoxetine nightly for one week. Atomoxetine dose will then be increased to 1.2 mg/kg/day (max 80 mg). During the low dose ato-oxy period, participants will take 5 mg oxybutynin and 0.5mg/kg/day (max 40 mg) atomoxetine. Dosing of the study treatment will occur approximately 30 minutes prior to bedtime. Participants who withdraw from the study will not be replaced.

Study participants will undergo eligibility screening that will include an initial screening to determine whether non- PSG enrollment criteria are met, followed by a 1 night in-lab PSG and health-related quality of life assessment for participants who qualify based on non-PSG criteria. For participants who are eligible and enroll in the study, the screening PSG night will serve as the baseline measure for apnea hypopnea index (AHI) and other PSG endpoints. On the final night of dosing for both high dose ato-oxy and low-dose ato-oxy, participants will return for inpatient PSG and health-related quality of life assessment. The primary efficacy endpoint is the change in obstructive AHI from baseline (high dose ato-oxy vs. low dose ato-oxy).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants between 6 to 17 years of age, inclusive, at the Screening Visit. Enrollment will be stratified to ensure equal representation of children age 6-12 and age 13-17. No more than 14 subjects will be randomized for each age group.
2. Known diagnosis of Down syndrome (trisomy 21, but not translocation or mosaicism)

Exclusion Criteria:

1. Hypoxemia independent of respiratory events on polysomnography (≥5 minutes with oxygen saturation <90%)
2. Presence of central sleep apnea on polysomnography (central AHI ≥ 5)
3. Currently using and adherent to PAP therapy (>4 hours per night for 70% of nights in the past 30 days based on device download or parent report)
4. MAO inhibitor use
5. Urinary retention
6. Prematurity < 37 weeks estimated gestational age
7. Seizure disorder
8. Untreated or inadequately treated hypothyroidism
9. Significant traumatic brain injury
10. Congenital heart disease and not cleared to participate by the patient's cardiologist
11. History of current, untreated depression
12. History of liver disease
13. 3+ or greater tonsillar hypertrophy.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Combs, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Combs D, Edgin J, Hsu CH, Bottrill K, Van Vorce H, Gerken B, Matloff D, La Rue S, Parthasarathy S. The combination of atomoxetine and oxybutynin for the treatment of obstructive sleep apnea in children with Down syndrome. J Clin Sleep Med. 2023 Dec 1;19(12):2065-2073. doi: 10.5664/jcsm.10764. PMID 37555595

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment was only 15 randomized participants rather than planned 24 due to recruitment delays related to the COVID-19 pandemic. 22 participants were enrolled but 7 did not qualify for randomization. 4 did not meet the requirement for apnea-hypopnea index >5 on their baseline polysomnogram, 1 had hypoxemia unrelated to OSA on their baseline polysomnogram, 1 could not tolerate polysomnogram and 1 participant became adherent to CPAP between consent and baseline polysomnogram.
Groups:
- High Dose Ato-oxy Then Low Dose Ato-oxy; Low Dose Ato-oxy Then High Dose Ato-oxy: Atomoxetine and oxybutynin (ato-oxy): Low dose ato-oxy will include 0.5 mg/kg/day of atomoxetine (max 40 mg) in combination with 5 mg oxybutynin High dose ato-oxy will include 1.2 mg/kg/day atomoxetine (max 80 mg) and 5 mg oxybutynin
Period: First Intervention
Arm/Group | High Dose Ato-oxy Then Low Dose Ato-oxy | Low Dose Ato-oxy Then High Dose Ato-oxy
Started | 8 | 7
Completed | 7 | 6
Not Completed | 1 | 1
Period: Second Intervention
Arm/Group | High Dose Ato-oxy Then Low Dose Ato-oxy | Low Dose Ato-oxy Then High Dose Ato-oxy
Started | 7 | 6
Completed | 7 | 5
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: Only participants with complete data were included in analysis. One participant did not have usable data on their final sleep study and is not included in these results.
Groups:
- All Study Participants: Atomoxetine and oxybutynin (ato-oxy): Low dose ato-oxy will include 0.5 mg/kg/day of atomoxetine (max 40 mg) in combination with 5 mg oxybutynin High dose ato-oxy will include 1.2 mg/kg/day atomoxetine (max 80 mg) and 5 mg oxybutynin
Arm/Group | All Study Participants
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.4 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
BMI percentile [Mean (Standard Deviation); unit: percentile] | 79 (23)
Congenital heart disease [Count of Participants; unit: Participants] | 8

OUTCOME MEASURES:

1. Primary Outcome: Obstructive Apnea-hypopnea Index (oAHI)
Description: change in number of obstructive apneas and hypopneas per hour on polysomnography from baseline
Time Frame: four weeks
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | High Dose Ato-oxy | Low Dose Ato-oxy
Number analyzed (Participants) | 11 | 11
events per hour | -3.79 (2.74) | -3.51 (3.06)

2. Secondary Outcome: Obstructive Sleep Apnea-18 Score (OSA-18)
Description: Change in OSA-18 (a measure of health-related quality of life) from baseline. The OSA-18 score ranges from 18 to 136, with lower scores indicating better health-related quality of life.
Time Frame: four weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose Ato-oxy | Low Dose Ato-oxy
Number analyzed (Participants) | 11 | 11
score on a scale | -6.00 (21.2) | -6.82 (11.91)

3. Secondary Outcome: Arousal Index
Description: change in number of arousals per hour on polysomnography from baseline
Time Frame: four weeks
Measure: Mean (Standard Deviation); unit: arousals per hour
Arm/Group | High Dose Ato-oxy | Low Dose Ato-oxy
Number analyzed (Participants) | 11 | 11
arousals per hour | 0.68 (8.24) | 2.01 (5.15)

4. Other Pre Specified Outcome: Pediatric Quality of Life Inventory (PedsQL) Total Score
Description: Change in PedsQL total score (a measure of health-related quality of life) from baseline. The PedsQL score ranges from 0-100, with higher scores indicating better health-related quality of life.
Time Frame: four weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose Ato-oxy | Low Dose Ato-oxy
Number analyzed (Participants) | 11 | 11
score on a scale | 1.97 (15.77) | 3.36 (15.27)

5. Other Pre Specified Outcome: Caregiver Global Impression of Change
Description: Change in Caregiver Global Impression of Change from baseline. This will be assessed on a seven point scale answering the question: Since the start of this therapy, my child's overall status is: 1. Very much improved; 2. Much improved; 3. Minimally Improved; 4. No change; 5. Minimally worse; 6. Much worse or 7. Very much worse.
Time Frame: four weeks
Population: Form not completed by one participant for high dose.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose Ato-oxy | Low Dose Ato-oxy
Number analyzed (Participants) | 10 | 11
score on a scale | 3.70 (0.95) | 3.45 (1.03)

6. Other Pre Specified Outcome: N1 Sleep Percentage
Description: Change in N1 sleep percentage on polysomnography from baseline
Time Frame: four weeks
Measure: Mean (Standard Deviation); unit: percentage of N1 sleep
Arm/Group | High Dose Ato-oxy | Low Dose Ato-oxy
Number analyzed (Participants) | 11 | 11
percentage of N1 sleep | 0.45 (3.49) | 0.40 (3.17)

7. Other Pre Specified Outcome: REM Sleep Percentage
Description: Change in REM sleep percentage on polysomnography from baseline
Time Frame: four weeks
Measure: Mean (Standard Deviation); unit: percentage of REM sleep
Arm/Group | High Dose Ato-oxy | Low Dose Ato-oxy
Number analyzed (Participants) | 11 | 11
percentage of REM sleep | -2.16 (10.16) | -1.41 (8.89)

8. Other Pre Specified Outcome: N3 Sleep Percentage
Description: Change in N3 sleep percentage on polysomnography from baseline
Time Frame: four weeks
Measure: Mean (Standard Deviation); unit: percentage of N3 sleep
Arm/Group | High Dose Ato-oxy | Low Dose Ato-oxy
Number analyzed (Participants) | 11 | 11
percentage of N3 sleep | -0.73 (14.58) | -4.29 (13.14)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout time on therapy (1 month each for high and low dose ato-oxy)
Description: Adverse events were assessed via weekly phone calls while on medications
Arm/Group | High Dose Ato-oxy | Low Dose Ato-oxy
All-Cause Mortality (participants affected / at risk) | 1/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/14
Other Adverse Events (participants affected / at risk) | 8/14 | 8/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Ato-oxy (N=14) | Low Dose Ato-oxy (N=14)
Respiratory failure and death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — One participant developed sepsis, respiratory failure and death while on high-dose ato-oxy. This appeared related to infectious cause and did not appear related to the study on DSMB review.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose Ato-oxy (N=14) | Low Dose Ato-oxy (N=14)
Fatigue (Psychiatric disorders) | 4 | 2
Mood changes (Psychiatric disorders) | 4 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 1
Headaches (Nervous system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Decreased urinary frequency (Renal and urinary disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT04115878/Prot_SAP_000.pdf